CLINICAL TRIAL: NCT03878147
Title: Culture-Specific Neurodevelopmental Assessment of HIV-affected Children
Brief Title: Neurodevelopmental Assessment of Children in Uganda and Malawi Using a Software Package
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other); Johns Hopkins University (Other); MU-JHU CARE (Other); Kamuzu University of Health Sciences (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael J. Boivin, Professor of Psychiatry and Neurology and Oftalmology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2191; R01HD098027 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: BPG Intervention; Control
Keywords: cognitive games, attention, memory, learning, reasoning, planning, HIV, African, children

STUDY DESIGN:
Intervention Model Description: The subject population for this proposal will consist of 600 children roughly equally divided between males and females and between HIV exposed uninfected and HIV unexposed and uninfected. These are Ugandan and Malawian children 5-12 years of age at study initiation who live in Uganda or Malawi.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BPG, Uganda (Experimental): Children in Uganda randomized to BPG
  Interventions: Behavioral: Cognitive Games Training
- Waitlist control, Uganda (No Intervention): Children in Uganda randomized to waitlist control
- BPG, Malawi (Experimental): Children in Malawi randomized to BPG
  Interventions: Behavioral: Cognitive Games Training
- Waitlist control, Malawi (No Intervention): Children in Malawi randomized to waitlist control

INTERVENTIONS:
Behavioral: Cognitive Games Training — Brain Powered Games (BPG) uses games for neurocognitive assessment and training, using images and sounds more familiar to African children. As a computerized cognitive rehabilitation training (CCRT) program designed for Sub-Saharan African school-age children, it can help children infected affected directly or indirectly by HIV. BPG consists of 5 core games evaluating different cognitive abilities (learning, memory, language, attention). Each game includes a visual tutorial, several adjustable settings on the administrative side (Admin), and records game play data for research purposes. Village Builder (VB) is a pro-social reasoning/planning world building strategy type game intended to evaluate frontal lobe executive functions in a culture-friendly and enjoyable game manner. It consists of many of the village artistic components as used in BPG but orchestrated into a village setting where children must gather resources and protect them in order to expand the capacity of the village.
  Other Names: Brain Powered Games; Village Builder
  Arms: BPG, Malawi; BPG, Uganda

SUMMARY:
The investigators will use Brain Power Games as a neurocognitive "stress test" or medical "challenge" test, in order to evaluate or improve brain/behavior functional integrity in HIV-affected children. This dual use of BPG is a key innovative feature. Each of the 5 core BPG games lasts 10 minutes and trains fine motor, monitoring/attention, visual/auditory working memory, spatial navigational learning.

The investigator's central hypothesis is that the BPG performance gains will be improved compared to waitlist control for children in Uganda and Malawi.

DETAILED DESCRIPTION:
We randomize equal numbers of each of three exposure groups of children (perinatally HIV infected, perinatally HIV-exposed but not infected, and unexposed/uninfected children) to one of two intervention arms. They are randomized to either the Brain Powered Games (BPG) intervention arm of 12 sessions of hour-long training (twice a day for several days weekly at the study clinic), or to the "wait-listed" arm of no BPG training sessions.

Separate analyses by country (Uganda and Malawi) are planned. HIV exposure status is used for balancing of randomization.

ELIGIBILITY:
Inclusion Criteria:

* HEU and HUU children at least 5 yrs of age and older from the PROMISE ND study (Uganda and Malawi)
* HIV+ children from P1104s (Uganda and Malawi)
* HUU children age-matched from PROMISE ND and P1104s study cohorts (Uganda and Malawi)

Exclusion Criteria:

* Medical history of serious birth complications
* Severe malnutrition
* Bacterial meningitis
* Encephalitis
* Cerebral malaria
* Other known brain injury or disorder requiring hospitalization
* Seizures or other neurological disabilities

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 599 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Johns Hopkins Research Project, Blantyre, Malawi
- Makerere University Johns Hopkins University Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
No individual-level data will be made available to other researchers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified by HIV exposure status (infected, exposed uninfected, unexposed uninfected) to ensure the same distribution of HIV exposure by trial arm (BPG or waitlist control). The study hypotheses were based on comparisons of BPG versus waitlist control arm across all children separately in Uganda and Malawi.
Period: Overall Study
Arm/Group | BPG, Uganda | Waitlist Control, Uganda | BPG, Malawi | Waitlist Control, Malawi
Started | 149 | 150 | 149 | 151
Completed | 146 | 146 | 147 | 149
Not Completed | 3 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Children In Uganda or Malawi aged 5-12 years
Groups:
- Total: Total of all reporting groups
Arm/Group | BPG, Uganda | Waitlist Control, Uganda | BPG, Malawi | Waitlist Control, Malawi | Total
Number analyzed (Participants) | 149 | 150 | 149 | 151 | 599
Age, Continuous [Mean (Standard Deviation); unit: years] — Child age in years
  years | 8.71 (2.41) | 9.01 (2.33) | 8.87 (2.12) | 9.03 (2.30) | 8.95 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 76 | 82 | 75 | 304
  Male | 78 | 74 | 67 | 76 | 295
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 149 | 150 | 149 | 151 | 599
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 0 | 0 | 149 | 151 | 300
  Uganda | 149 | 150 | 0 | 0 | 299
HIV status [Count of Participants; unit: Participants]
  HIV unexposed uninfected | 59 | 61 | 61 | 59 | 240
  HIV exposed uninfected | 60 | 59 | 59 | 61 | 239
  HIV infected | 30 | 30 | 29 | 31 | 120
Kaufman Assessment Battery for Children 2nd Edition (KABC-II) Mental Processing Index (MPI) [Mean (Standard Deviation); unit: units on a scale] — The KABC mental processing index (MPI) is a summary score across domains. The normative mean of 100 and standard deviation of 15 are based on American norms. Higher score is better.
  units on a scale | 71.54 (9.83) | 71.65 (11.05) | 70.47 (10.03) | 68.82 (11.59) | 69.64 (10.86)
Test of Variables of Attention (TOVA) attention deficit hyperactivity disorder (ADHD) index [Mean (Standard Deviation); unit: units on a scale] — TOVA is a computerized visual continuous performance test used in to screen, diagnose and monitor children and adults at risk for ADHD. TOVA consists of the rapid (tachistoscopic) presentation of a large geometric square on the computer screen with a smaller dark box either in the upper position (signal) or lower position (non-signal). The child is asked to press a switch in response to the signal (measuring vigilance attention), but to withhold responding to the non-signal (measuring impulsivity). The potential range of the TOVA ADHD index is from -10 to 10, higher score is better.
  units on a scale | -1.72 (3.12) | -1.50 (2.96) | -3.14 (3.30) | -3.16 (3.10) | -3.15 (3.20)
Cognitive State (CogState) correct moves per second [Mean (Standard Deviation); unit: number of moves per second] — CogState presents a 30-min session that includes playing cards in a game-like manner to assess memory, attention, discrimination learning, and executive function that is non-language dependent. The number of correct moves per second during maze learning reflects executive functioning/planning. Higher number reflects better outcome.
  number of moves per second | 0.13 (0.10) | 0.15 (0.09) | 0.14 (0.17) | 0.16 (0.20) | 0.15 (0.18)

OUTCOME MEASURES:

1. Primary Outcome: Kaufman Assessment Battery for Children 2nd Edition (KABC-II) Mental Processing Index (MPI)
Description: The KABC mental processing index (MPI) is a summary score across domains. The normative mean 100 and standard deviation 15 are based on American norms. Range is 43 to 160. Higher score reflects better outcome.
Time Frame: Month 2, month 6
Population: Children in Uganda and Malawi
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BPG, Uganda | Waitlist Control, Uganda | BPG, Malawi | Waitlist Control, Malawi
Number analyzed (Participants) | 149 | 150 | 149 | 151
units on a scale
  Month 2 | 77.18 (0.60) | 74.79 (0.61) | 71.79 (0.71) | 73.72 (0.72)
  Month 6 | 77.27 (0.60) | 76.46 (0.61) | 73.40 (0.69) | 73.61 (0.70)
Statistical Analysis 1: Comparison: BPG, Uganda vs Waitlist Control, Uganda; The null hypothesis was that the means of two arms were equal. The alternative hypothesis was that means of two arms were not equal. With this sample size, differences between arms corresponding to the unadjusted effect size Cohen's d=0.33 would be detectable as statistically significant with power of .80 in two-sided tests at .05 level of significance; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p < .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = 2.39, 95% CI 2-sided [0.78 to 4.01], Standard Error of Mean 0.82 — BPG minus waitlist control
Statistical Analysis 2: Comparison: BPG, Uganda vs Waitlist Control, Uganda; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 6; p = .32, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.80 to 2.44], Standard Error of Mean 0.82 — BPG minus waitlist control
Statistical Analysis 3: Comparison: BPG, Malawi vs Waitlist Control, Malawi; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p = .07, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-3.74 to 0.16], Standard Error of Mean 0.99 — BPG minus waitlist control
Statistical Analysis 4: Comparison: BPG, Malawi vs Waitlist Control, Malawi; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 6; p = .83, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-2.10 to 1.68], Standard Error of Mean 0.96 — BPG minus waitlist control

2. Secondary Outcome: Test of Variables of Attention (TOVA) Attention Deficit Hyperactivity Disorder (ADHD) Index
Description: TOVA is a computerized visual continuous performance test used in to screen, diagnose and monitor children and adults at risk for ADHD. TOVA consists of the rapid (tachistoscopic) presentation of a large geometric square on the computer screen with a smaller dark box either in the upper position (signal) or lower position (non-signal). The child is asked to press a switch in response to the signal (measuring vigilance attention), but to withhold responding to the non-signal (measuring impulsivity). The potential range of the TOVA ADHD index is from -10 to 10, higher score is better.
Time Frame: Month 2, month 6
Population: Children in Uganda and Malawi.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | BPG, Uganda | Waitlist Control, Uganda | BPG, Malawi | Waitlist Control, Malawi
Number analyzed (Participants) | 149 | 150 | 149 | 151
units on a scale
  Month 2 | -1.21 (0.21) | -1.08 (0.21) | -2.63 (0.25) | -2.35 (0.25)
  Month 6 | -0.81 (0.21) | -0.83 (0.21) | -2.23 (0.24) | -2.15 (0.24)
Statistical Analysis 1: Comparison: BPG, Uganda vs Waitlist Control, Uganda; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p = .65, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.71 to 0.42], Standard Error of Mean 0.28 — BPG minus waitlist control
Statistical Analysis 2: Comparison: BPG, Uganda vs Waitlist Control, Uganda; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 6; p = .95, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Median Difference (Final Values) = 0.02, 95% CI 2-sided [-0.54 to 0.58], Standard Error of Mean 0.29 — BPG minus waitlist control
Statistical Analysis 3: Comparison: BPG, Malawi vs Waitlist Control, Malawi; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p = .34, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Median Difference (Final Values) = -0.39, 95% CI 2-sided [-0.92 to 0.13], Standard Error of Mean 0.27 — BPG minus waitlist control
Statistical Analysis 4: Comparison: BPG, Malawi vs Waitlist Control, Malawi; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 6; p = .81, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.73 to 0.58], Standard Error of Mean 0.33 — BPG minus waitlist control

3. Secondary Outcome: Cognitive State (CogState) Correct Moves Per Second
Description: CogState presents a 30-minute session that includes playing cards in a game-like manner to assess memory, attention, discrimination learning, and executive function that is non-language dependent. The number of correct moves per second during maze learning reflects executive functioning/planning. The range is from 0 to 5. Higher number reflects better outcome.
Time Frame: Month 2, month 6
Population: Children in Uganda and Malawi.
Measure: Least Squares Mean (Standard Error); unit: moves per second
Arm/Group | BPG, Uganda | Waitlist Control, Uganda | BPG, Malawi | Waitlist Control, Malawi
Number analyzed (Participants) | 149 | 150 | 149 | 151
moves per second
  Month 2 | 0.23 (0.01) | 0.21 (0.01) | 0.20 (0.01) | 0.18 (0.01)
  Month 6 | 0.27 (0.01) | 0.25 (0.01) | 0.23 (0.01) | 0.22 (0.01)
Statistical Analysis 1: Comparison: BPG, Uganda vs Waitlist Control, Uganda; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p = .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Median Difference (Final Values) = 0.02, 95% CI 2-sided [0.004 to 0.043], Standard Error of Mean 0.01 — BPG minus waitlist control
Statistical Analysis 2: Comparison: BPG, Uganda vs Waitlist Control, Uganda; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 6; p = .02, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [0.003 to 0.040], Standard Error of Mean 0.01 — BPG minus waitlist control
Statistical Analysis 3: Comparison: BPG, Malawi vs Waitlist Control, Malawi; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p = .19, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 0.05], Standard Error of Mean 0.01 — BPG minus waitlist control
Statistical Analysis 4: Comparison: BPG, Malawi vs Waitlist Control, Malawi; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was difference between least square means of trial arms at month 2; p = .19, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. A priori threshold for statistical significance was .05; Baseline value of the outcome, child's age, sex, and HIV exposure status were included as covariates; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.01 to 0.04], Standard Error of Mean 0.01 — BPG minus waitlist control

ADVERSE EVENTS:
Time Frame: Adverse even data were collected over 6 months of study participation for all children.
Arm/Group | BPG, Uganda | Waitlist Control, Uganda | BPG, Malawi | Waitlist Control, Malawi
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/150 | 0/149 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/150 | 0/149 | 0/151
Other Adverse Events (participants affected / at risk) | 0/149 | 0/150 | 0/149 | 0/151

LIMITATIONS AND CAVEATS:
There were multiple secondary outcomes with no formal adjustment for the level of significance. The results for the primary outcome should be given greatest strength of the interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03878147/Prot_SAP_ICF_000.pdf